CLINICAL TRIAL: NCT05095857
Title: S-ketamine for Cortical Spreading Depolarisation in Patients With Severe Acute Brain Injury
Brief Title: The Anaesthetic Ketamine as Treatment for Patients With Severe Acute Brain Injury
Acronym: KETA-BID
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Trine Hjorslev Andreasen, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21056972; 2021-003716-12 (EudraCT Number)
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Intracerebral Hemorrhage; Traumatic Brain Injury
Keywords: Cortical Spreading Depolarisation; Ketamine
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage; Brain Injuries, Traumatic | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-ketamine (Active Comparator): S-ketamine is given as a continuous infusion started at a dose of 2.0 mg/kg/hour. The infusion rate will be re-evaluated after 24 hours, where (1) the infusion will be stopped if 24 hours ensue without SDs, (2) maintained at 2.0 mg/kg/hour if the 24-hour incidence of SDs decreases below the rate of the previous 24 hours but SD is not totally abolished, or (3) increased to 3.0 mg/kg/hour if the incidence of SD is at or above the rate of the previous 24 hours. If the infusion rate has been increased to 3.0 mg/kg/hour, the rate will be returned to 2.0 mg/kg/hour if 24 consecutive hours of ECoG show no SD.
  Interventions: Drug: S-ketamine
- Isotonic saline (Placebo Comparator): Isotonic saline is given as placebo. It will be given as a continuous infusion started at a dose corresponding to a dose of S-ketamine of 2.0 mg/kg/hour, and follow the criteria for increasing/decreasing infusion rates as S-ketamine. The infusion rate is read from a table listing different infusion rates (ml/hour) based on participant weight and if the treatment tier corresponds to a S-ketamine dose of 2 or 3 mg/kg/hour.
  Interventions: Other: Isotonic saline (placebo)

INTERVENTIONS:
Drug: S-ketamine — S-ketamines is an NMDA-receptor antagonist with sedative and analgesic properties. It will in the present trial be given in sedative doses (2-3 mg/kg/hour) in case of clustered SDs following a dosing algorithm according to SD occurrence.
  Other Names: Esketamine
  Arms: S-ketamine
Other: Isotonic saline (placebo) — Isotonic saline has the same appearance as S-ketamine with both being clear liquids with no bubbles or other distinguishing features.
  Arms: Isotonic saline

SUMMARY:
Cortical spreading depolarisations are pathological depolarisation waves that occur frequently after severe acute brain injury and has been associated with poor outcome. S-ketamine has been shown to inhibit cortical spreading depolarisations. The aim of the present study is to examine the efficacy and safety of using S-ketamine for treatment of patients with severe acute brain injury, as well as the feasibility of the trial design.

DETAILED DESCRIPTION:
Severe acute brain injury caused by traumatic brain injury (TBI), aneurysmal subarachnoid haemorrhage (aSAH) or intracerebral haemorrhage (ICH) carries a high morbidity and mortality. In all these conditions, clinical neurological deterioration may occur as a consequence of so-called secondary brain injury, which reduces the chance of a good outcome. Thus, neurological deterioration after the initial injury is generally associated with a worse outcome. Cortical spreading depolarisations (SDs) are pathological depolarisation waves that occur frequently after both TBI, SAH, and ICH and have been related to poor outcome. The SDs, which can be detected by electrocorticography (ECoG, using electrodes placed directly on the brain cortex), propagate across the cerebral cortex and are followed by an excessive upregulation of cerebral metabolism and decrease in cerebral blood flow. In vulnerable brain tissue such as in patients after acute primary brain injury, this combination of hypermetabolism and hypoperfusion is thought to increase the risk of ischaemia and infarction. The anaesthetic drug ketamine, which is an NMDA-receptor antagonist, appears to inhibit SDs both in vitro and in patient series.

The present trial is a randomised, blinded, placebo-controlled, parallel-group pilot and feasibility trial, where participants with clustered SD despite physiological optimisation are allocated 1:1 to infusion of S-ketamine versus matching placebo. In the present trial, participants admitted to the neurointensive care unit with TBI, aSAH or ICH and undergoing craniotomy or craniectomy (for clipping of an aneurysm or removal of a space-occupying haematoma). Patients are monitored at the neurointensive care unit, Rigshospitalet and sedated using standard sedatives. Patients will be monitored both with ECoG, intracranial pressure (ICP), brain tissue oxygen tension (PbtO2), and microdialysis. Patients in whom SDs occur will be subjected to a protocol of physiological optimisation targeting ICP, PbtO2, blood glucose and core temperature following clinical guidelines. If clustered SDs occur despite optimisation, patients are randomly allocated to infusion of either S-ketamine or matching placebo (isotonic saline) at a 1:1 allocation ratio with full blinding of the treatment allocation.

The present trial will continue until 160 participants have been randomised. Since only participants with clustered SDs are randomised, the investigators expect to include no more than 400 participants for ECoG monitoring.

The present trial aims to examine the efficacy of S-ketamine on SDs, the safety, and the feasibility of the trial design. Furthermore, surviving patients will be followed up until six months after the injury, and functional outcome will be recorded by the modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Admitted to the NICU with a diagnosis of traumatic brain injury (TBI), aneurysmal subarachnoid haemorrhage (aSAH) or spontaneous intracerebral haemorrhage (ICH).
* Planned for surgery with a supratentorial craniotomy or craniectomy.
* Expected to continue sedation and mechanical ventilation after surgery.

Exclusion Criteria:

* Neither patient or next of kin understand Danish or English.
* Known allergy to S-ketamine (the active pharmaceutical ingredient or the excipients).
* Wake-up call to occur immediately after surgery.
* Pregnancy (all female participants aged ≤ 50 years will have a urine or blood hCG taken to control for pregnancy).
* Active anti-psychotic treatment before admission.
* Current abuse of ketamine.
* Decision to withdraw active treatment.
* ICH secondary to a known brain tumour at the time of inclusion.

Since this is an emergency trial informed consent will be obtained from a trial guardian before inclusion of the participant, and informed consent will be sought from next of kin as soon as possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of SDs after randomisation | From randomisation to end of ECoG monitoring, expected to be a maximum of 14 days
  Efficacy of S-ketamine on the occurrence of cortical spreading depolarisations

SECONDARY OUTCOMES:
Rate of adverse events and adverse reactions | During treatment with S-ketamine or placebo, a maximum of 14 days
Functional outcome at 6 months after randomisation | 6 months after randomisation
  assessed using modified Rankin Scale

OTHER OUTCOMES:
All-cause mortality | assessed at 6 months after randomisation
Number of participants with signs of ischaemia or infarction on computed tomography (CT) or magnetic resonance imaging (MRI). | Before discharge from NICU or the semi-intentisive care unit, expected up to be no later than day 21 postrandomisation
  Last scan performed on clinical indication before discharge from NICU or semi-intensive care unit
Occurrence of metabolic crisis (defined as microdialysis (MD)-lactate/pyruvate ratio >40, MD-glucose < 0.8 μmol/L) | Postrandomisation period, expected up to 21 days
Occurrence of local cerebral hypoxia (PbtO2 <20 mmHg for more than 20 minutes) | Postrandomisation period, expected up to 21 days
Dosage of standard sedatives and analgesics | Postrandomisation period, expected up to 21 days
Number of imaging procedures (CT of the brain, CT-angiography, digital subtraction angiography, MRI) | Postrandomisation period, expected up to 21 days
Number of episodes of neurological worsening | Postrandomisation period, expected up to 21 days
Occurrence of delayed cerebral ischemia (DCI) in participants with aSAH | Postrandomisation period, expected up to 21 days
Fraction of participants included in the trial out of all eligible participants | Assessed after 2 years or when one-third of the 160 participants have been randomised
  Feasibility outcome
Fraction of participants who are randomised of all included | Assessed after 2 years or when one-third of the 160 participants have been randomised
  Feasibility outcome

CONTACTS AND LOCATIONS:
Overall Officials: Trine H Andreasen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Macdonald RL, Schweizer TA. Spontaneous subarachnoid haemorrhage. Lancet. 2017 Feb 11;389(10069):655-666. doi: 10.1016/S0140-6736(16)30668-7. Epub 2016 Sep 13. PMID 27637674
- [Background] Nieuwkamp DJ, Setz LE, Algra A, Linn FH, de Rooij NK, Rinkel GJ. Changes in case fatality of aneurysmal subarachnoid haemorrhage over time, according to age, sex, and region: a meta-analysis. Lancet Neurol. 2009 Jul;8(7):635-42. doi: 10.1016/S1474-4422(09)70126-7. Epub 2009 Jun 6. PMID 19501022
- [Background] Zhou YT, Tong DM, Wang SD, Ye S, Xu BW, Yang CX. Acute spontaneous intracerebral hemorrhage and traumatic brain injury are the most common causes of critical illness in the ICU and have high early mortality. BMC Neurol. 2018 Aug 27;18(1):127. doi: 10.1186/s12883-018-1127-z. PMID 30149796
- [Background] Gross BA, Jankowitz BT, Friedlander RM. Cerebral Intraparenchymal Hemorrhage: A Review. JAMA. 2019 Apr 2;321(13):1295-1303. doi: 10.1001/jama.2019.2413. PMID 30938800
- [Background] Gruenbaum SE, Zlotnik A, Gruenbaum BF, Hersey D, Bilotta F. Pharmacologic Neuroprotection for Functional Outcomes After Traumatic Brain Injury: A Systematic Review of the Clinical Literature. CNS Drugs. 2016 Sep;30(9):791-806. doi: 10.1007/s40263-016-0355-2. PMID 27339615
- [Background] Gruenbaum SE, Bilotta F. Postoperative ICU management of patients after subarachnoid hemorrhage. Curr Opin Anaesthesiol. 2014 Oct;27(5):489-93. doi: 10.1097/ACO.0000000000000111. PMID 25115766
- [Background] Seder DB, Mayer SA. Critical care management of subarachnoid hemorrhage and ischemic stroke. Clin Chest Med. 2009 Mar;30(1):103-22, viii-ix. doi: 10.1016/j.ccm.2008.11.004. PMID 19186283
- [Background] Sheriff FG, Hinson HE. Pathophysiology and clinical management of moderate and severe traumatic brain injury in the ICU. Semin Neurol. 2015 Feb;35(1):42-9. doi: 10.1055/s-0035-1544238. Epub 2015 Feb 25. PMID 25714866
- [Background] Shah S, Kimberly WT. Today's Approach to Treating Brain Swelling in the Neuro Intensive Care Unit. Semin Neurol. 2016 Dec;36(6):502-507. doi: 10.1055/s-0036-1592109. Epub 2016 Dec 1. PMID 27907954
- [Background] Gradisek P, Osredkar J, Korsic M, Kremzar B. Multiple indicators model of long-term mortality in traumatic brain injury. Brain Inj. 2012;26(12):1472-81. doi: 10.3109/02699052.2012.694567. Epub 2012 Jun 21. PMID 22721420
- [Background] Olsen MH, Orre M, Leisner ACW, Rasmussen R, Bache S, Welling KL, Eskesen V, Moller K. Delayed cerebral ischaemia in patients with aneurysmal subarachnoid haemorrhage: Functional outcome and long-term mortality. Acta Anaesthesiol Scand. 2019 Oct;63(9):1191-1199. doi: 10.1111/aas.13412. Epub 2019 Jun 7. PMID 31173342
- [Background] Cordonnier C, Demchuk A, Ziai W, Anderson CS. Intracerebral haemorrhage: current approaches to acute management. Lancet. 2018 Oct 6;392(10154):1257-1268. doi: 10.1016/S0140-6736(18)31878-6. PMID 30319113
- [Background] Budohoski KP, Guilfoyle M, Helmy A, Huuskonen T, Czosnyka M, Kirollos R, Menon DK, Pickard JD, Kirkpatrick PJ. The pathophysiology and treatment of delayed cerebral ischaemia following subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2014 Dec;85(12):1343-53. doi: 10.1136/jnnp-2014-307711. Epub 2014 May 20. PMID 24847164
- [Background] Lauritzen M, Dreier JP, Fabricius M, Hartings JA, Graf R, Strong AJ. Clinical relevance of cortical spreading depression in neurological disorders: migraine, malignant stroke, subarachnoid and intracranial hemorrhage, and traumatic brain injury. J Cereb Blood Flow Metab. 2011 Jan;31(1):17-35. doi: 10.1038/jcbfm.2010.191. Epub 2010 Nov 3. PMID 21045864
- [Background] Hartings JA, Andaluz N, Bullock MR, Hinzman JM, Mathern B, Pahl C, Puccio A, Shutter LA, Strong AJ, Vagal A, Wilson JA, Dreier JP, Ngwenya LB, Foreman B, Pahren L, Lingsma H, Okonkwo DO. Prognostic Value of Spreading Depolarizations in Patients With Severe Traumatic Brain Injury. JAMA Neurol. 2020 Apr 1;77(4):489-499. doi: 10.1001/jamaneurol.2019.4476. PMID 31886870
- [Background] Helbok R, Schiefecker AJ, Friberg C, Beer R, Kofler M, Rhomberg P, Unterberger I, Gizewski E, Hauerberg J, Moller K, Lackner P, Broessner G, Pfausler B, Ortler M, Thome C, Schmutzhard E, Fabricius M. Spreading depolarizations in patients with spontaneous intracerebral hemorrhage: Association with perihematomal edema progression. J Cereb Blood Flow Metab. 2017 May;37(5):1871-1882. doi: 10.1177/0271678X16651269. Epub 2016 Jan 1. PMID 27207168
- [Background] Dreier JP, Woitzik J, Fabricius M, Bhatia R, Major S, Drenckhahn C, Lehmann TN, Sarrafzadeh A, Willumsen L, Hartings JA, Sakowitz OW, Seemann JH, Thieme A, Lauritzen M, Strong AJ. Delayed ischaemic neurological deficits after subarachnoid haemorrhage are associated with clusters of spreading depolarizations. Brain. 2006 Dec;129(Pt 12):3224-37. doi: 10.1093/brain/awl297. Epub 2006 Oct 25. PMID 17067993
- [Background] Ayata C, Lauritzen M. Spreading Depression, Spreading Depolarizations, and the Cerebral Vasculature. Physiol Rev. 2015 Jul;95(3):953-93. doi: 10.1152/physrev.00027.2014. PMID 26133935
- [Background] Chesnut RM, Marshall LF, Klauber MR, Blunt BA, Baldwin N, Eisenberg HM, Jane JA, Marmarou A, Foulkes MA. The role of secondary brain injury in determining outcome from severe head injury. J Trauma. 1993 Feb;34(2):216-22. doi: 10.1097/00005373-199302000-00006. PMID 8459458
- [Background] Welling L, Welling MS, Teixeira MJ, Figueiredo EG. Cortical spread depolarization and ketamine: a revival of an old drug or a new era of neuroprotective drugs? World Neurosurg. 2015 Apr;83(4):396-7. doi: 10.1016/j.wneu.2015.01.006. Epub 2015 Jan 31. No abstract available. PMID 25644895
- [Background] Reinhart KM, Shuttleworth CW. Ketamine reduces deleterious consequences of spreading depolarizations. Exp Neurol. 2018 Jul;305:121-128. doi: 10.1016/j.expneurol.2018.04.007. Epub 2018 Apr 10. PMID 29653188
- [Background] Sakowitz OW, Kiening KL, Krajewski KL, Sarrafzadeh AS, Fabricius M, Strong AJ, Unterberg AW, Dreier JP. Preliminary evidence that ketamine inhibits spreading depolarizations in acute human brain injury. Stroke. 2009 Aug;40(8):e519-22. doi: 10.1161/STROKEAHA.109.549303. Epub 2009 Jun 11. PMID 19520992
- [Background] Hertle DN, Dreier JP, Woitzik J, Hartings JA, Bullock R, Okonkwo DO, Shutter LA, Vidgeon S, Strong AJ, Kowoll C, Dohmen C, Diedler J, Veltkamp R, Bruckner T, Unterberg AW, Sakowitz OW; Cooperative Study of Brain Injury Depolarizations (COSBID). Effect of analgesics and sedatives on the occurrence of spreading depolarizations accompanying acute brain injury. Brain. 2012 Aug;135(Pt 8):2390-8. doi: 10.1093/brain/aws152. Epub 2012 Jun 19. PMID 22719001
- [Background] Schiefecker AJ, Beer R, Pfausler B, Lackner P, Broessner G, Unterberger I, Sohm F, Mulino M, Thome C, Humpel C, Schmutzhard E, Helbok R. Clusters of cortical spreading depolarizations in a patient with intracerebral hemorrhage: a multimodal neuromonitoring study. Neurocrit Care. 2015 Apr;22(2):293-8. doi: 10.1007/s12028-014-0050-4. PMID 25142825
- [Background] Hertle DN, Heer M, Santos E, Scholl M, Kowoll CM, Dohmen C, Diedler J, Veltkamp R, Graf R, Unterberg AW, Sakowitz OW. Changes in electrocorticographic beta frequency components precede spreading depolarization in patients with acute brain injury. Clin Neurophysiol. 2016 Jul;127(7):2661-7. doi: 10.1016/j.clinph.2016.04.026. Epub 2016 May 4. PMID 27291885
- [Background] Carlson AP, Abbas M, Alunday RL, Qeadan F, Shuttleworth CW. Spreading depolarization in acute brain injury inhibited by ketamine: a prospective, randomized, multiple crossover trial. J Neurosurg. 2018 May 25;130(5):1513-1519. doi: 10.3171/2017.12.JNS171665. Print 2019 May 1. PMID 29799344
- [Derived] Andreasen TH, Olsen MH, Gluud C, Lindschou J, Fabricius M, Hauerberg J, Moller K. S-ketamine versus placebo for cortical spreading depolarisation in severe acute brain injury (KETA-BID): protocol for a pilot, randomised, blinded clinical trial. BMJ Open. 2025 Jul 28;15(7):e101426. doi: 10.1136/bmjopen-2025-101426. PMID 40721263